CLINICAL TRIAL: NCT04416321
Title: A Prospective, Non-comparative, Single-centre, Post-market Clinical Study to Evaluate the Safety and Performance of PEEK-OPTIMA™ HA Enhanced Interbody Cages for the Treatment of Degenerative Disc Disease in the Lumbar Spine
Brief Title: A Clinical Study to Evaluate Safety and Performance of PEEK-OPTIMA™ HA Enhanced.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Invibio Ltd (Industry)
Collaborators: Keos LLC (Unknown); Medical Metrics Diagnostics, Inc (Industry); Technomics Research (Industry); Viedoc Technologies (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KEOS01
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2025-04

CONDITIONS: Degenerative Disc Disease; Spondylolisthesis; Retrolisthesis
Keywords: Lumbar Degenerative Disc Disease; Spondylolisthesis; retrolisthesis
MeSH Terms: conditions — Intervertebral Disc Degeneration; Spondylolisthesis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Intervention Model Description: All subjects recruited and will receive the Keos Lumbar Interbody Fusion Device
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Device (Other): All subjects who are entered into this trial will receive the Keos Lumbar Interbody Fusion Device.
  Interventions: Device: Surgery with the Keos Lumbar Interbody Fusion Device

INTERVENTIONS:
Device: Surgery with the Keos Lumbar Interbody Fusion Device — All subjects will received the Keos Lumbar Interbody Fusion Device if according to the investigators opinion they are clinically indicated to have surgery treatment for degenerative disc disease, spondylolisthesis and retrolisthesis

SUMMARY:
The purpose of this trial is to collect clinical outcomes including radiographic and CT outcomes in patients who undergo spinal fusion using the Keos Lumbar Interbody Fusion Device.

DETAILED DESCRIPTION:
This prospective, non-comparative, single-center, post-market trial will evaluate the safety and efficacy of the PEEK-OPTIMA ™ HA Enhanced Keos Lumbar Interbody Fusion Device in patients suffering from degenerative disc disease, spondylolisthesis and retrolisthesis in the lumbar spine. The trial will capture clinical outcomes, radiographic and CT outcomes over a 24 month period post operatively. One centre will be involved in the recruitment of 30 patients the clinic involved will focus on this type of treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years of age or older.
2. Primary diagnosis of symptomatic degenerative disc disease (DDD) or symptomatic degenerative disc disease (DDD) with spondylolisthesis (Grade 1), or retrolisthesis, at one or two contiguous levels from L2 to S1.
3. Have discogenic back pain.
4. Suitable for transforaminal lumbar interbody fusion (TLIF) surgery.
5. Indicated for surgical treatment with the Keos Lumbar IBFD with autologous bone graft.
6. Completed at least 6 months of conservative non-operative treatment.
7. Female subjects of childbearing age must have a negative pregnancy test.
8. Able to understand this clinical study, co-operate with procedures.
9. Able to give voluntary, written informed consent to participate.

Exclusion Criteria:

1. Not undergone previous spinal surgery at the affected disc level(s).
2. Evidence of tumour and/or malignant disease.
3. Known osteoporosis or severe osteopenia.
4. Known rheumatoid arthritis, ankylosing spondylitis or who are immunocompromised.
5. Known allergy to the material used in the instrumentation.
6. Evidence of an active infection.
7. Any conditions outlined as contraindicated in the Instructions for Use.
8. Receiving any drug treatment that may affect bone metabolism.
9. Female subjects who are pregnant or lactating.
10. Current smokers or have stopped smoking less than 6 months ago.
11. Known drug or alcohol abusers.
12. Currently enrolled in a clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-01-27 (Actual); Study Completion 2026-01-27 (Actual)

PRIMARY OUTCOMES:
Interbody fusion rate | 6 months post - operatively
  Interbody fusion will be graded along the superior and inferior interfaces separately in 25% increments

SECONDARY OUTCOMES:
To measure how much pain the subject is in according to a pain scale 0-10 | 6 weeks, 3, 6, 12 and 24 months post operatively
  Visual analogue scale for back and leg 0-10 cm (no pain - worst possible pain)
To measure the Quality of Life of the subject according to a set list of questions: Questionnaire SF-12 | pre-operatively, 6 weeks, 3, 6, 12 and 24 months post operatively
  Questionnaire SF-12 collection of questions health related to assess vitality, physical functioning, bodily pain, general health perceptions, emotional and physical functioning, social and mental health. Patients will pick from a set list of answers for each health related question. The responses on each item are scored and summarised into Physical and Mental Health Composite Scores (PCS & MCS) and range from 0-100. The lower the score the more disability. The higher the score the less disability i.e.a score of zero is equivalent to maximum disability and a score of 100 is equivalent to no disability.
Functional Impairment | pre-operatively, 6 weeks, 3, 6, 12 and 24 months post operatively
  Questionnaire ODI (Oswestry Disability Index) - disability questionnaire used to assess functional impairment of the patient. Regarding lifting, ability to walk, sit, stand, sleep, travel and graded by score of 0-100 (0= no disability and 100= maximum disability possible)

CONTACTS AND LOCATIONS:
Overall Officials: Louis A Marotti, M.D. PhD, Principal Investigator — Neurosurgical Associates of Lancaster
Locations (1):
- Neurosurgical Associates of Lancaster, Lancaster, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No